CLINICAL TRIAL: NCT03430648
Title: Is Tau Protein Linked to Mobility Function?
Acronym: SYNERGY
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00042050; P30AG021332 (NIH)
Record Dates: First submitted 2018-02-05; First posted 2018-02-13 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease; Physical Activity
Keywords: Tau protein; PET imaging; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Motor Activity; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cognitively and metabolically normal: This group has been defined as being cognitively and metabolically normal.
- Cognitively normal with prediabetes: This group has been defined as being cognitively normal but showing signs of prediabetes.
- Persons with Mild Cognitive Impairment: This group has been defined as being mildly cognitively impaired.
- Persons with early Alzheimer's disase: This group has been defined as having early Alzheimer's disease.

SUMMARY:
This project will provide new data to address an important question linking Alzheimer's disease neuropathology to physical disability.

DETAILED DESCRIPTION:
Impaired mobility is strongly linked to cognitive function and vice versa. Cognitive functions are strongly associated with mobility function, most commonly assessed using gait speed. In the Health ABC Study, Digit Symbol Substitution Test (DSST) and Modified Mini Mental Status (3MS) scores were significantly associated with gait speed and gait speed decline. Poor lower extremity performance predicts faster age-related cognitive decline and increased incidence of mild cognitive impairment (MCI) and dementia. This study will explore the role of tau protein as the neuropathologic basis for these associations.

Brain imaging markers may be the link between cognitive measures and gait. White matter disease is commonly measured by quantifying white matter (WM) lesion load, which is associated with small vessel ischemic disease. More subtle microstructural changes can be observed by calculating fractional anisotropy (FA) from diffusion tensor imaging (DTI). Aging is accompanied by changes in cortical volume, white matter microstructure and an increased prevalence of WM lesions. WM lesions have been strongly implicated in declining physical function. These brain changes are associated with impaired balance, slower movement speeds, slower chair stand times and increased falls risk.Recently, Aâ accumulation in the brain has also been linked to slow gait. This finding suggests a pathologic mechanism linking Alzheimer s disease processes to gait impairments. However, Aâ accumulation itself may not be the critical neuropathic change. In recent studies of Aâ42 and phosphorylated tau protein in cerebral spinal fluid, it has been found that low Aâ42 levels themselves are not associated with impaired cognition, but that elevated tau levels are also required. If the process of cognitive impairment parallels the process of gait impairment, it might be that tau levels are more important correlates of gait changes. To the investigators' knowledge the relationship between CSF tau levels and mobility has never been explored. PET ligands for brain tau have recently become available, but the relationship between brain tau accumulation and gait has yet to be determined. In this study, investigators will relate gait characteristics to CSF Aâ42 and phosphorylated tau levels, and perform brain PET imaging in a subset to related tau protein accumulation to gait characteristics for the first time. Both mobility impairment and Alzheimers disease (AD) occur in the context of the aging vascular system. Over the past 15 years, it has been recognized that abnormalities of thoracic aortic stiffness are associated with the development of abnormalities in small vessels supplying the brain and kidneys. As the aorta stiffens, the propagation speed of the systolic flow wave increases through the aortic lumen. (Stiffness within the thoracic aorta can be accomplished through measurement of aortic pulse wave velocity.) In hypertensive patients, aortic archway pulse wave velocity has been associated with increases in left ventricular mass as well as lacunar brain infarcts independent of age, sex, and the duration of hypertension. In the Multi-Ethnic Dallas Heart Study aortic arch pulse wave velocity is an independent predictor of white matter hyper-intensities. In those with diabetes, increasing aortic stiffness contributes to the development of small vessel microvascular dysfunction which is associated with deep white matter atrophy as well as cognitive decline. Recently, a stiffness mismatch between the thoracic aorta and small vessels within the cerebral microcirculation has been described. This mismatch impacts microvascular pulsatility and appears to diminish diffusion anisotrophy between the cerebral spinal fluid and the CNS microcirculation. This observation may contribute to retained amyloid type protein in those with AD.

ELIGIBILITY:
Inclusion Criteria:

* 50+ years of age and participated in the Wake Forest Alzheimer's Disease Core Center study
* Willing to provide informed consent
* Not dependent on a walker

Exclusion Criteria:

* Recent cardiac event in the last 6 months
* Uncontrolled hypertension (BP >200/110 mmHg)
* Neurological (e.g., Parkinson's) or hematological disease
* Participants with a knee replacement in last 6 months
* Participants with recent eye surgery in last 6 months
* Severe musculoskeletal impairment (e.g., sciatica, fibromyalgia, severe leg/back pain)
* If willing to get an MRI, must not have indwelling metal-contraining prosthesis, pacemaker or defibrillator, history of welding, permanent make up or head/neck tattoo, or any other contraindication to MRI

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators plan to recruit a total of 60 people age 50 and older from the Wake Forest Alzheimer's Disease Research Center's Clinical Core group.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Association between CSF total and phosphorylated tau levels and gait speed | Baseline
  This will be done using the 400m walk test.
Association between CSF total and phosphorylated tau levels and gait variability | Baseline
  This will be done using the gaitrite mat.
Association between CSF total and phosphorylated tau levels and standing balance. | Baseline
  This will be done using the AMTI force plate.

SECONDARY OUTCOMES:
Examine the association between Digit Symbol Substitution Test and gait speed | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kritchevsky, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States